CLINICAL TRIAL: NCT06599619
Title: A Study of the Effects of Anti-PD1 Adjuvant Checkpoint Blockade Immunotherapy on Features of Atypical/Dysplastic Nevi in Patients With Stage IIB-IIIC Melanoma
Brief Title: Effects of Anti-PD1 Adjuvant Checkpoint Blockade Immunotherapy on Atypical/Dysplastic Nevi
Status: Recruiting | Type: Observational
Sponsor: John Kirkwood (Other)
Collaborators: Melanoma Research Foundation (Other); VeyTel Inc. (Unknown)
Responsible Party: Sponsor-Investigator, John Kirkwood, Professor of Medicine, Immunology, and Dermatology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: HCC 23-167
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Melanoma
Keywords: anti-PD1 therapy; immune checkpoint blockade; dysplastic nevi; BRAF and NRAS mutations
MeSH Terms: conditions — Melanoma; Dysplastic Nevus Syndrome; Hereditary Sensory and Autonomic Neuropathies | interventions — Pharmaceutical Preparations; Nivolumab; pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy of one nevus will be performed at baseline (A) and at 3 month follow up (B). Tissue biopsies will be obtained after photographs and dermoscopic imaging has been performed at each time point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Treated with single agent, adjuvant anti-PD1 therapy: Patients receiving single agent, adjuvant anti-PD1 therapy (given either as standard of care or as part of a separate investigational study)
  Interventions: Drug: Single agent, adjuvant anti-PD1 therapy

INTERVENTIONS:
Drug: Single agent, adjuvant anti-PD1 therapy — One of the following Single-agent, adjuvant anti-PD1 therapies:
  Nivolumab is a type of targeted therapy drug called an immune checkpoint inhibitor (a type of immunotherapy). It is a monoclonal antibody that binds to the protein PD-1 on the surface of immune cells called T cells. It works by keeping cancer cells from suppressing the immune system.
  Dose = 240 mg IV every 2 weeks/480 mg every 4 weeks or, Pembrolizumab is a monoclonal antibody and a type of immune checkpoint inhibitor that's used in cancer immunotherapy. It works by attaching to the PD-1 protein on the surface of T cells, which are immune cells. This prevents cancer cells from suppressing the immune system, allowing the immune system to attack and kill the cancer cells.
  Dose = 200 mg IV every 3 weeks/ 400 mg every 6 weeks
  Other Names: OPDIVO®; Keytruda; Pembrolizumab; Nivolumab

SUMMARY:
This study will examine the impact of anti-programmed cell death 1 (PD1) therapy given in the approved adjuvant therapeutic regimens upon the morphologic, histopathologic, molecular and immunologic as well as genomic features of atypical/dysplastic nevi (A/DN) in patients with a prior documented melanoma of Stages IIB, IIC, IIIA, IIIB, or IIIC and concurrent presence of two or more atypical nevi.

DETAILED DESCRIPTION:
Given the established efficacy of anti-PD1 therapy as an adjuvant treatment in both advanced nodal and earlier stage deep primary node negative melanoma, this study hypothesizes that anti-PD1 therapy may provide a basis for effective therapeutic prevention. To study if anti-PD1 therapy can help prevent the development of melanoma, this study will examine its effects upon atypical/dysplastic nevi, which are well established as non-obligate pre-cursor lesions that are markers of increased risk of melanoma. This single agent, adjuvant study will evaluate the impact of adjuvant anti-PD1 therapy on morphology, histopathology, immunologic/molecular features, and gene expression of atypical/dysplastic nevi present in patients with stage IIB-III melanoma. This study aims to determine if anti-PD1 therapy will increase CD8 T cell responses to melanoma antigens, resulting in immune surveillance and anti-tumor immune responses within A/DN. It postulates that in response to anti-PD1 therapy, the aggregate pigmentation of total nevi including atypical/dysplastic nevi and benign melanocytic nevi will decrease with a measurable morphologic response. This study also asserts that there will be histopathologic changes within A/DN including increased density of immune infiltrate and increased presence of regression features. Increased anti-tumor immune response measured by increased CD8, IFN-y, and PD-1 expression within nevi is anticipated, along with a decrease in genes involved in pathways of melanomagenesis, pigmentation, and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have at least two atypical nevi of ≥ 4 mm diameter.
2. Subjects must have a current documented history of melanoma.
3. Subject must be ≥ 18 years and if female of childbearing potential, must agree to practice effective contraception per institutional SOC if sexually active.
4. Subjects will have been deemed candidates for adjuvant therapy with single agent anti-PD1 therapy.
5. Subjects must give written informed consent to participate in this study with consent signed and dated prior to entry into trial.

Exclusion Criteria:

1. Patients with non-malignant diseases or indications that would preclude the administration of anti-PD1 therapy such as significant immune suppression or active autoimmune disease requiring disease modifying, immunosuppressive therapy, will be ineligible.
2. Patients who have previously received anti-PD1 therapy
3. Patients with history of other active, non-melanoma cancers
4. Patients who are receiving other anti-neoplastic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a prior documented melanoma of Stages IIB, IIC, IIIA, IIIB, or IIIC and concurrent presence of two or more atypical nevi who have received anti-programmed cell death 1 (PD1) therapy given in the approved adjuvant therapeutic regimens.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Change in the aggregate pigmentation | Pre-treatment, up to 12 months
  Percentage change in the total aggregate pigmentation including A/DN and benign melanocytic nevi. Percent change will be quantified from posterior trunk digital photographic images utilizing DermViz automated image comparison software.

SECONDARY OUTCOMES:
Change in predefined atypical nevi - size | Pre-treatment, up to 12 months
  Change in size of predefined atypical nevi at the level of the individual nevus, as documented by dermoscopy. An expert clinician panel will evaluate pre- and post-treatment dermoscopic images in a blinded manner to score the visual features of nevus atypia.
Change in predefined atypical nevi - margin | Pre-treatment, up to 12 months
  Change in margin of predefined atypical nevi at the level of the individual nevus, as documented by dermoscopy. An expert clinician panel will evaluate pre- and post-treatment dermoscopic images in a blinded manner to score the visual features of nevus atypia.
Change in predefined atypical nevi - pigmentation | Pre-treatment, up to 12 months
  Change in pigmentation of predefined atypical nevi at the level of the individual nevus, as documented by dermoscopy. An expert clinician panel will evaluate pre- and post-treatment dermoscopic images in a blinded manner to score the visual features of nevus atypia.
Change in histopathologic features of A/DN - cellular infiltrate | Pre-treatment, up to 12 months
  Histopathologic changes within atypical nevi that are biopsied will be assessed by an expert dermatopathologist for the dendritic cell and lymphocytic cell immune infiltrate.
Change in histopathologic features of A/DN - regression features | Pre-treatment, up to 12 months
  Histopathologic changes within atypical nevi that are biopsied will be assessed by an expert dermatopathologist for regression features including fibrosis and vascularization.
Change in histopathologic features of A/DN - cytologic features | Pre-treatment, up to 12 months
  Histopathologic changes within atypical nevi that are biopsied will be assessed by an expert dermatopathologist for cytologic features including nuclear size and atypia.
Change in histopathologic features of A/DN - dysplastic features | Pre-treatment, up to 12 months
  Histopathologic changes within atypical nevi that are biopsied will be assessed by an expert dermatopathologist for dysplastic features of nevi including cell architecture.

OTHER OUTCOMES:
Change in Expression of SOX-10 and BRAF | Pre-treatment, up to 12 months
  Quantify change in expression of key genes of melanomagenesis in A/DN in response to anti-PD1 therapy, measured via bulk RNA-sequencing performed on biopsied nevus specimens.
Change in CD-8 T lymphocytes | Pre-treatment, up to 12 months
  Changes in the immune microenvironment of A/DN in response to anti-PD1 therapy. Changes in T cell subsets will be quantified and compared pre- and post-treatment via multiplex IHC and multiplex IF performed on biopsied specimens.
Change in T-regs | Pre-treatment, up to 12 months
  Changes in the immune microenvironment of A/DN in response to anti-PD1 therapy. Changes in regulatory T cells will be quantified and compared pre- and post-treatment via multiplex IHC and multiplex IF performed on biopsied specimens.
Change in IFN-y immune transcriptional signature | Pre-treatment, up to 12 months
  Changes in the immune microenvironment of A/DN in response to anti-PD1 therapy. Changes in IFN-y immune transcriptional signature will be quantified and compared pre- and post-treatment via multiplex IHC and multiplex IF performed on biopsied specimens.
Change in IL-6 immune transcriptional signature | Pre-treatment, up to 12 months
  Changes in the immune microenvironment of A/DN in response to anti-PD1 therapy. Changes in Immune transcriptional signature will be quantified and compared pre- and post-treatment via multiplex IHC and multiplex IF performed on biopsied specimens.
Change in IL-10 immune transcriptional signature | Pre-treatment, up to 12 months
  Changes in the immune microenvironment of A/DN in response to anti-PD1 therapy. IL-10 immune transcriptional signature will be quantified and compared pre- and post-treatment via multiplex IHC and multiplex IF performed on biopsied specimens.
Change in PD1 expression | Pre-treatment, up to 12 months
  Changes in the immune microenvironment of A/DN in response to anti-PD1 therapy. Changes in PD1 expression will be quantified and compared pre- and post-treatment via multiplex IHC and multiplex IF performed on biopsied specimens.

CONTACTS AND LOCATIONS:
Overall Officials: John M Kirkwood, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No